CLINICAL TRIAL: NCT03065491
Title: Effect of Red Yeast Rice, Phytosterols and L-tyrosol on Lipid Profile and Endothelial Function: a Double-blind, Placebo-controlled, Randomized Clinical Trial
Brief Title: Effect of Red Yeast Rice, Phytosterols and L-tyrosol on Lipid Profile and Endothelial Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Claudio Borghi, Principal Investigator, Professor Claudio Borghi, University of Bologna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MPT_trial_2016
Record Dates: First submitted 2017-02-15; First posted 2017-02-28 (Actual); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Hypercholesterolemia
Keywords: Red yeast rice; Phytosterols; L-Tyrosol; Lipids; LDL-cholesterol; Endothelial function
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active treatment (Active Comparator): Combined nutraceutical
  Interventions: Dietary Supplement: Combined nutraceutical
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Combined nutraceutical — Plant sterols 800 mg + Red Yeast Rice containing 5 mg monacolin K + L-Tyrosol 50 mg per daily dose Oral administration: 1 tablet per day
  Arms: Active treatment
Other: Placebo — Oral administration: 1 tablet per day
  Arms: Placebo

SUMMARY:
A large body of evidence confirm the cholesterol lowering effect of red yeast rice, phytosterols and L-tyrosol. Because their mechanisms of action mime the ones of chemical statins and cholesterol absorption inhibitors, it is plausible that their association will provide a more relevant (and safe) LDL cholesterolemia reduction.

DETAILED DESCRIPTION:
European Food Safety Authority approves some health claim related to the cardiometabolic effects of some nutraceuticals, and in particular of red yeast rice, phytosterols and L-tyrosol.

In a previous study the investigators have already demonstrated the synergistic effect of red yeast rice and phytosterols in term of lipid-lowering activity.

Preliminary data suggest that these nutraceuticals could also exert a positive effect on vascular health beyond the direct effects on serum lipids.

No data are available on the combined effects of these dietary supplement in humans.

ELIGIBILITY:
Inclusion Criteria:

* Suboptimal LDL level (115-160 mg/dL)
* TG<400 mg/dL
* Signed informed consent form

Exclusion Criteria:

* Patients already affected by cardiovascular diseases (secondary prevention) or with estimated 10 years cardiovascular disease risk> 10 years
* LDL-C<115 mg/dL or >160 mg/dL, TG>400 mg/dL
* Obesity (BMI>30 kg/m2) or diabetes mellitus
* Assumption of lipid lowering drugs or dietary supplements, or drugs potentially affecting the lipid metabolism
* Antihypertensive treatment not stabilized since at least 3 months
* Known current thyroid, gastrointestinal or liver diseases
* Any medical or surgical condition that would limit the patient adhesion to the study protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2017-02-17 (Actual)

PRIMARY OUTCOMES:
LDL-cholesterolemia absolute reduction from baseline and between groups | 8 weeks
  Absolute reduction of LDL-cholesterolemia after 8 weeks of treatment
LDL-cholesterolemia % reduction from baseline and between groups | 8 weeks
  % reduction of LDL-cholesterolemia after 8 weeks of treatment

SECONDARY OUTCOMES:
Flow-mediated dilation improvement from baseline and between groups | 8 weeks
  % vascular heath improvement after 8 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Borghi, MD, Principal Investigator — S. Orsola-Malpighi University Hospital
Locations (1):
- S. Orsola-Malpighi University Hospital, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No